CLINICAL TRIAL: NCT03231683
Title: The Use of S+Ketamine Versus Placebo During Target-Controlled Intravenous Anaesthesia to Reduce Morphine Consumption and Side Effects After Abdominal Hysterectomy: A Randomized Controlled Trial
Brief Title: Use of S+Ketamine During Target-Controlled Intravenous Anaesthesia After Abdominal Hysterectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EC 200801014
Record Dates: First submitted 2015-09-03; First posted 2017-07-27 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2016-09

CONDITIONS: Ketamine; Anesthesia; Morphine; Hysterectomy
MeSH Terms: interventions — Esketamine; Ketamine; Sodium Chloride; Remifentanil; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Esketamine (Active Comparator): Esketamine and remifentanil to be given alongside with propofol through target control infusion pump.
  Interventions: Drug: Esketamine; Drug: Remifentanil; Drug: Propofol
- Control (Placebo Comparator): Saline and remifentanil to be given alongside with propofol through target control infusion pump.
  Interventions: Drug: Saline; Drug: Remifentanil; Drug: Propofol

INTERVENTIONS:
Drug: Esketamine — intravenous S+ketamine 0.25 mg/kg (i.v. bolus) at the beginning and 0.25 mg/kg (i.v. bolus) 20 minutes before extubation along with remifentanil according to Minto model and propofol according to Marsh model
  Other Names: S+ ketamine
  Arms: Esketamine
Drug: Saline — intravenous normal saline (as placebo, with similar volume) at the beginning and 20 minutes before extubation along with remifentanil according to Minto model and propofol according to Schnider model
  Other Names: Sodium chloride
  Arms: Control
Drug: Remifentanil — Either S+ketamine or saline at the beginning and 20 minutes before extubation along with remifentanil according to Minto model and propofol according to Schnider model
  Other Names: Ultiva
Drug: Propofol — Either S+ketamine or saline at the beginning and 20 minutes before extubation along with remifentanil according to Minto model and propofol according to Schnider model
  Other Names: Diprivan

SUMMARY:
The investigators want to investigate the effect of low dose S+ ketamine compared to placebo on cumulative morphine consumption at 24 hours in 90 women undergoing open abdominal hysterectomy with remifentanil-propofol target controlled infusion (TCI) in KK Women's and Children's Hospital. The secondary aims are to investigate the use of low dose S+ ketamine on the incidence of nausea, vomiting, pruritus (opioid side effect), sedation score and psycho mimetic assessment compared to placebo group. The investigators propose to conduct a double blinded, randomized controlled study in women undergoing open abdominal hysterectomy with remifentanil-propofol TCI. (1) Treatment Group: intravenous ketamine 0.5 mg/kg at the beginning and 0.5 mg/kg 20 minutes before extubation. (2) Control Group: intravenous normal saline (as placebo) at the beginning and 20 minutes before extubation.

DETAILED DESCRIPTION:
A number of 90 American Society of Anesthesiologists (ASA) I and II patients undergoing elective open abdominal hysterectomies will be randomly distributed in two groups of 45 patient's each and assigned to receive one of the of the following:

1. Treatment Group: intravenous S+ketamine 0.25 mg/kg (i.v. bolus) at the beginning and 0.25 mg/kg (i.v. bolus) 20 minutes before extubation along with remifentanil according to Minto model and propofol infusion according to Marsh model through target control infusion pump.
2. Control Group: intravenous normal saline (as placebo, with similar volume) at the beginning and 20 minutes before extubation along with remifentanil according to Minto model and propofol according to Schnider model through target control infusion pump.

Randomization procedure is performed by the unblinded study team investigator. Patients will be randomized to either the treatment or control groups with a 1:1 allocation ratio. Sequence generation will be performed using a computerized random number generator, employing a permuted block randomization scheme. Allocation concealment will be maintained by having the random numbers pre-generated by an off-site statistician who will not be involved in subject recruitment. Implementation will be via serially numbered opaque sealed envelopes.

Throughout the study period, blinded study members will perform drug administration and data collection, while unblinded study members will be in charge for the investigational drug storage, dispensing and preparation. Any premature unblinding (e.g. accidental unblinding, unblinding due a serious adverse event) of the investigational product will be promptly documented and explained. In the case of adverse effect or severe adverse effect requiring information on the study treatment to manage a patient, the treatment code of the patient will be unblinded.

ELIGIBILITY:
Inclusion Criteria:

* Female ASA I/II patients above age of 21 years old scheduled gynecological open surgery for benign condition (fibroids, adenomyosis), who are willing and able to give written informed consent for participation in this study.

Exclusion Criteria:

* Contraindications to the use of S+ ketamine, as listed in the product label e.g. untreated or insufficiently treated thyroid hyperfunction, unstable angina pectoris or myocardial infarction within the last 6 months, diseases of the central nervous system, increased intraocular pressure and perforating ocular injuries, surgical procedures in the upper respiratory tract;
* History of drug or alcohol abuse;
* Regular use of analgesics, or use of opioids within 12 hours of surgery;
* Chronic use of benzodiazepine or neuroleptics;
* Thyroid replacement hormone;
* History of ischaemic heart disease, hypertension, psychiatric disorder;
* BMI> 30kg/m2;
* Laparoscopic surgery converted to open surgery;
* Pregnant or breast feeding females.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Post-operative Cumulative morphine consumption at 24 hours | 1 day
  Post-operative Cumulative morphine consumption at 24 hours will be measured in the S-ketamine group compared to the placebo group

SECONDARY OUTCOMES:
Incidence of nausea | 1 day
  The use of low dose S-ketamine will reduce the incidence of nausea / vomiting, pruritus (opioid side effect) compared to placebo in women undergoing open abdominal hysterectomy with remifentanil-propofol target controlled infusion.
Incidence of vomiting | 1 day
  The use of low dose S-ketamine will reduce the incidence of nausea / vomiting, pruritus (opioid side effect) compared to placebo in women undergoing open abdominal hysterectomy with remifentanil-propofol target controlled infusion.
Incidence of pruritus | 1 day
  The use of low dose S-ketamine will reduce the incidence of nausea / vomiting, pruritus (opioid side effect) compared to placebo in women undergoing open abdominal hysterectomy with remifentanil-propofol target controlled infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Farida Ithnin, MBBCh, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- Kk Women'S and Children'S Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No